CLINICAL TRIAL: NCT03812094
Title: The Efficacy of Basic Bladder Advice and Alarm Therapy in Nocturnal Enuresis - a Randomized Controlled Trial
Brief Title: Basic Bladder Advice and Alarm Therapy in Nocturnal Enuresis
Acronym: BAAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalarna County Council, Sweden (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Barbro Hedin Skogman, MD, associate professor, Dalarna County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAAT-01
Record Dates: First submitted 2019-01-07; First posted 2019-01-22 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Nocturnal Enuresis
Keywords: paediatric, children, treatment, intervention
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trail
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Basic Bladder advice (Active Comparator): Basic bladder advice as given from a pre-specified document, study nurse
  Interventions: Behavioral: Basic Bladder advice
- Alarm (Active Comparator): Alarm Enurad 400
  Interventions: Device: Enurad 400
- No treatment (No Intervention): No treatment during study period.

INTERVENTIONS:
Device: Enurad 400 — Alarm treatment
  Arms: Alarm
Behavioral: Basic Bladder advice — Pre-specified Basic bladder advice
  Arms: Basic Bladder advice

SUMMARY:
Enuresis is the scientific term for bedwetting. Modern research has established three pathogenic mechanisms as crucial:

1. Excessive urine production at night (nocturnal polyuria).
2. Detrusor over activity. The bladder may contract regardless of whether it is full or not.
3. Difficulties to arouse from sleep and will not wake up when the bladder is full or contracts.

Children with daytime incontinence usually suffer from detrusor over activity and many of them are constipated. The reason for this connection is probably partly anatomical; constipated children have to use the rectum as a storage space, and the chronically distended rectum will compress the bladder from behind.

The link between constipation and enuresis (as opposed to daytime incontinence) is less clear although it is logically plausible. Our experience is that some enuretic children become dry at night just by treatment of constipation, but this is yet not supported by sufficient evidence The standard primary treatment of enuresis - as reflected by global consensus guidelines - rests upon three pillars. The recommended first step is 1) bladder advice. The next step, if the child is still wet at night, is either 2) the antidiuretic drug desmopressin or 3) the sleep-modifying enuresis alarm.

The underlying idea behind basic bladder advice is that the child is taught to more actively take command over the bladder by voiding according to a regular daytime schedule, using correct voiding posture and spread fluid intake evenly across the day. The rationale behind the recommendation of this strategy is that is the established cornerstone of the treatment of daytime incontinence and that detrusor over activity is a pathogenic factor common to both conditions. By influencing bladder, function during the day it is assumed that nocturnal bladder function will also normalize. The problem is a glaring lack of evidence.

Our primary aims with this study is to better understand which roles basic bladder advice, constipation therapy and/or the enuresis alarm play in the first-line therapy of enuresis.

DETAILED DESCRIPTION:
Treatment strategies in nocturnal enuresis

BACKGROUND. Enuresis is the scientific term for bedwetting. Approximately one in ten children in early school age suffers from this condition. Modern research has established three pathogenic mechanisms as crucial:

1. Excessive urine production at night (nocturnal polyuria). The bladder is filled to capacity before the night is over.
2. Nocturnal detrusor overactivity. In these cases, the bladder may contract regardless of whether it is full or not.
3. Almost all children with enuresis are difficult to arouse from sleep and will not wake up when the bladder is full or contracts.

Regardless of which of the above factors is relevant in the individual child, the condition is often inherited.

All enuretic children do not wet their beds every night, but even children who experience wet nights sporadically may be very much bothered by their condition - they may, for instance, not dare to participate in school camps or sleepovers. Many of the children also suffer from concomitant daytime incontinence.

Enuresis is not, as previously thought, primarily a psychiatric disorder. It has psychiatric consequences, but only rarely psychiatric causes. Enuretic children, as group, have lower self-esteem than their dry peers, and their quality of life is also negatively affected. Another link between the bladder and the psychological wellbeing of the child is that, for unclear reasons, enuresis (as well as daytime incontinence) is overrepresented among children with neuropsychiatric disturbances such as ADHD, and vice versa. These considerations make the successful treatment of enuresis extra important.

THE BLADDER-BOWEL LINK. It is well established that children with daytime incontinence usually suffer from underlying detrusor overactivity and that many of them are constipated. Treatment of daytime incontinence in these children will usually only be successful if the constipation is also treated. The reason for this connection is probably partly anatomical; constipated children have to use the rectum as a storage space, and the chronically distended rectum will compress the bladder from behind.

The link between constipation and enuresis (as opposed to daytime incontinence) is less clear although it is logically plausible. Our experience is that some enuretic children become dry at night just by treatment of constipation, but this is as yet not supported by sufficient evidence. We neither know how common constipation is among enuretic children, nor how important this, when present, is to treat.

CLINICAL EVALUATION OF THE ENURETIC CHILD. Children who seek medical attention for uncomplicated enuresis usually do not need any complicated or invasive evaluation. No blood samples need to be taken and no radiological or urodynamic examinations are motivated. A nurse with a basic knowledge of pediatric bladder problems best evaluates children. If you know how to ask, the right questions the very few children with enuresis due to serious underlying conditions will easily be found.

The bladder diary plays a crucial role in the evaluation of children with bladder problems. By writing down how often and how much urine the child voids during a few days, and by assessing nocturnal urine production via the weighing of diapers or sheet covers, important information is gained regarding bladder and kidney function during day and night. Additional relevant information is provided if the family documents wet and dry nights, as well as bowel movements, during two weeks.

TREATMENT. The standard primary treatment of enuresis - as reflected by global consensus guidelines - rests upon three pillars. The recommended first step is 1) bladder advice, or basic bladder advice. The next step, if the child is still wet at night, is either 2) the antidiuretic drug desmopressin or 3) the sleep-modifying enuresis alarm.

The underlying idea behind basic bladder advice is that the child is taught to take command over the bladder by voiding according to a regular day-time schedule, using correct voiding posture and spread fluid intake evenly across the day. The rationale behind the recommendation of this strategy is that is the established cornerstone of the treatment of daytime incontinence and that detrusor over activity is a pathogenic factor common to both conditions. By influencing bladder function during the day it is assumed that nocturnal bladder function will also normalize.

The problem is a glaring lack of evidence. We do not know that daytime bladder training has any influence at all on nocturnal enuresis. And the therapy, although completely harmless, demands lots of nursing time and family commitment. We recently performed the first ever randomised, controlled study of basic bladder advice in enuretic children and found no effect. However, these results need to be further explored and confirmed before we know if the global recommendations should be changed. Furthermore, during our completed study the therapy was given during four weeks only and all participating children suffered from frequent enuresis (i.e. enuresis occurring >50% of the nights). Thus, we still do not know whether the treatment will help if it is given during a longer period or if children with infrequent enuresis do have a beneficent effect of the therapy.

Desmopressin is taken at bedtime and, being an analogue to human vasopressin, decreases nocturnal urine production. It helps 30-50% of enuretic children to achieve dry nights as long as it is taken but has only limited, if any, curative effect.

The enuresis alarm is a device that gives off a strong alarm signal every time there is urine in the bed. The method is well-established and has a clearly curative effect in more than half of the children who use it, even though the therapeutic mechanism is slightly unclear. Presumably, the use of the alarm either influences sleep and arousal mechanisms so the child wakes up to void or learns to semi consciously inhibit nocturnal detrusor contractions; in both cases, the enuresis disappears. The main problem with the alarm is that it demands a high degree of motivation and compliance by the child and it may take months until full effect is achieved.

In spite of these strategies, many enuretic children, perhaps 25%, are therapy-resistant. For these children, who have experienced only failures, the burden and associated psychosocial risks are extra high.

PROGNOSTIC INDICATORS Since different enuretic children have different causes behind their bedwetting they will also respond differently to therapies. Much would be won if we could choose correct therapy for the individual child at the first try.

It is known that desmopressin is likely (although not certain) to be beneficial if the bladder diary shows that the nocturnal urine production is high and the daytime voided volumes (volumes per micturition) are normal. However, prognostic indicators for alarm response are much less studied - which is frustrating, given the high amount of work required for this therapy.

We may presume that family motivation and the ability to follow instructions are prognostically favourable indicators, but this assumption has never been properly tested. There are some studies indicating that the alarm works best for children with frequent enuresis but it is unclear whether factors such as nocturnal urine production, daytime micturition habits, or indeed anamnestic data, give any prognostic information.

From the above background, it is clear that there are several questions that need to be answered if a better, individualized and cost-effective enuresis therapy is to be achieved.

PRIMARY AIMS To better understand which roles basic bladder advise, constipation therapy and/or the enuresis alarm play in the first-line therapy of enuresis.

SECONDARY AIMS

* Is constipation more common among enuretic children than normal controls?
* In enuretic children with constipation, how large effect against the enuresis has treatment of the constipation?
* Do easily acquired data from the bladder diary give prognostic information as regarding the antienuretic effect of basic bladder training and/or the alarm?
* Do children with infrequent enuresis respond differently to therapy than those who wet their beds most nights?
* Which therapy is perceived as most cumbersome for the families - basic bladder advice or the enuresis alarm? METHODS PROJECT I - ENURESIS AND CONSTIPATION. All patients and controls visit the study nurse. They are asked a number of questions concerning bladder and bowel habits and undergo non-invasive urodynamic examination, i.e. they empty their bladder on the uroflow toilet and have any residual urine (urine left in the bladder after voiding) detected via ultrasound. Ultrasound is also used to assess the diameter of the rectum just behind the bladder. These procedures are all part of the routine evaluation of children with bladder issues and involve no violation of privacy.

The nurse then supplies the family with a bladder diary, which is to be completed at home. The following data is gathered:

* Wet and dry nights during two weeks (only patients)
* Nycturia (awake voiding's at night) during two weeks
* Voided volumes at each voiding during two days
* Fluid intake during two days and nights
* Weighing of diapers or sheet covers during three nights (only patients)
* Bowel movements during two weeks In addition to this the nurse notes the completeness of the data and how long it takes for the family to return the bladder diary; i.e. the family's motivation and ability to comply with the instructions is also assessed.

Enuretic children who have shown signs/symptoms of constipation (infrequent bowel movements, faecal incontinence or a rectal diameter >30 mm) will be given standard laxative therapy and their enuresis will be reassessed.

PROJECT II - RANDOMIZED COMPARISON BETWEEN BASIC UROTHERAPY, THE ENURESIS ALARM AND NO TREATMET All enuretic children who completed project I and still suffer from enuresis - including those who have been given treatment for constipation but did not become dry - will be invited to take part in the randomised study. The participants will be randomised into three groups. Regardless of group all children will be given information about bladder function and enuresis pathogenesis, and all ongoing laxative therapy will continue.

The children will be randomized in to tree groups, "basic bladder advise", "alarm" or "no treatment".

* Group A. Basic bladder advice is given in accordance with international guidelines. A qualified pediatric nurse/ urotherapist give the treatment during 8 weeks. Contact by phone is given in week 2 and 6. During the last two weeks (week 7 and 8) wet and dry nights are again documented. At the end of treatment the family grades the level of workload and disruption that the treatment has incurred.
* Group B. Alarm therapy according to international guidelines. Contact by phone is given after in week 2 and 6. During the last two weeks (week 7 and 8) wet and dry nights are again documented. At the end of treatment the family grades the level of workload and disruption that the treatment has incurred.
* Group C. These children are given no active treatment. During the last two week, 7 and 8 wet and dry nights are again documented.

Regardless of which therapy has been given (or not given) the children who still wet their beds after completion of project II will be given an appointment to the pediatric outpatient ward for further treatment.

IMPLICATIONS AND RELEVANCE Through the results of this project we believe that first-line treatment for a very large number of enuretic children will be improved, simplified and rationalized. The impact will be international and global treatment recommendations may be changed.

ELIGIBILITY:
Inclusion criteria:

* Children 6-11 Years
* Enuresis (monosymtomatic enuresis)

Exclusion criteria:

* Day incontinence (nonmonosymtomatic enuresis)
* Neurological disease
* Urological malformation
* Kidney disease
* Previous alarm treatment for enuresis
* Don´t want to stop medication whit Vasopressin (if currant)

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Reduction of wet nights per two weeks as compared to baseline enuresis frequency. | 14 days mesurement before study compered to 14 days in treatment week 7 and 8
  Respons to treatment is at least 3 nights per two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Malin Borgström, Study Director — Center for Clinical Research Dalarna
Locations (1):
- Center for Clinical Research Dalarna, Falun, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borgstrom M, Bergsten A, Tunebjer M, Hedin Skogman B, Neveus T. Daytime urotherapy in nocturnal enuresis: a randomised, controlled trial. Arch Dis Child. 2022 Jun;107(6):570-574. doi: 10.1136/archdischild-2021-323488. Epub 2022 Jan 24. PMID 35074830